CLINICAL TRIAL: NCT00048880
Title: Phase I Study of HeFi-1 in Refractory CD30-Positive Malignancy
Brief Title: Phase I Study of HeFi-1 to Treat Cancers With CD30 Protein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030038; 03-C-0038; NCT00053079 (obsolete NCT alias)
Record Dates: First submitted 2002-11-08; First posted 2002-11-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-03-05

CONDITIONS: Neoplasms
Keywords: Anaplastic Large Cell Lymphoma; Monoclonal Antibody; CD30; Antibody Saturation; Apoptosis; Flow Cytometry; Cancer
MeSH Terms: conditions — Neoplasms; Lymphoma, Large-Cell, Anaplastic

INTERVENTIONS:
Drug: HeFi-1 Monoclonal Antibody

SUMMARY:
Background:

* Some cancers, such as Hodgkin's disease, anaplastic large cell lymphoma and others, have a protein on the surface of the cancer cell called CD30.
* HeFi-1 is an antibody that binds to the CD30 protein and sends signals to the cancer cells that can cause them to die.

Objectives:

* To determine the highest dose of HeFi-1 that can safely be given to patients with tumors that have the CD30 protein.
* To determine the response of the tumor to treatment with HeFi-1.

Eligibility:

* Patients 18 years of age and older with Hodgkin's disease, anaplastic large cell lymphoma, cutaneous T cell lymphoma and adult T cell leukemia or lymphoma who have signs of tumor growth or recurrence following standard treatment
* Patients' tumor cells must have the CD30 protein.

Design:

* Groups of three patients are treated with increasingly higher doses of HeFi-1 (ranging from 0.5 to 5 mg/kg) to determine the highest safe dose.
* HeFi-1 is infused through a vein on 4 days, followed by 2 days of rest over a 10-day period. Patients may receive up to 2 treatment courses if they show some response and do not have severe side effects.
* Blood samples are collected several times during the study to determine safety. A lymph node biopsy is done at the beginning of the study to test the effect of HeFi-1 on cancer cells in the test tube, and a bone marrow biopsy may be done at the end of treatment if the bone marrow was positive for tumor cells at the beginning of treatment.

DETAILED DESCRIPTION:
BACKGROUND:

The scientific basis for this study is the observation that antibodies directed at the ligand-binding site of CD30 induce apoptosis in vitro and cure animals bearing CD30-positive tumors.

HeFi-1, a murine monoclonal antibody developed at the NCI, specifically binds human CD30, a member of the tumor necrosis receptor superfamily, at the ligand-binding site.

CD30 is expressed on activated T-cells, Reed-Sternberg cells, anaplastic large cell lymphoma, and some AIDS-related lymphoma cells.

Tumor cells from patients with anaplastic large cell lymphoma are sensitive to the effects of HeFi-1 but Hodgkin's disease cell lines show variable responsiveness due to the presence of mutations in I B kinase which result in constitutive activation of NF- B.

OBJECTIVE:

The primary objective of this study is to determine the toxicity and maximum tolerated dose of HeFi-1 in patients with CD30-positive malignancy.

This study will explore the pharmacokinetics, dose required to saturate CD30 binding sites in tumor aspirates, and the frequency and time course of onset of development of human anti-mouse antibody (HAMA).

These studies will allow us to monitor in a preliminary fashion the clinical tumor response, measured by reduction in tumor lesions and by following the tumor marker serum soluble interleukin 2 receptor.

ELIGIBILITY:

Patients with measurable or evaluable CD30-positive lymphoma who have become refractory to standard therapy, including Hodgkin's disease, systemic anaplastic large cell lymphoma, cutaneous T cell lymphoma and adult T cell leukemia/lymphoma are eligible for treatment.

DESIGN:

This is a phase I dose-escalation trial in which cohorts of three patients will be treated with HeFi-1 ranging from 0.5 to 5 mg/kg/dose (total dose of 2 to 20 mg/kg per treatment course).

Four doses will be given on an every three days schedule over a 10-day period for each cycle.

Two cycles of therapy will be administered provided the patient has had a partial or complete response and has not developed dose-limiting toxicity or HAMA.

ELIGIBILITY:
* INCLUSION CRITERIA:

All Patients must have a histologically confirmed diagnosis of malignancy by department of pathology at the enrolling institution.

Tumor cells must express CD30. CD30 expression will be verified by immunohistochemistry. At least 30% of tumor cells must be CD30 positive. CD30 staining will be performed on existing tissue blocks and on fresh tumor tissue if a biopsy is performed.

Patients must have measurable or evaluable disease.

The patient must have a granulocyte count of at least 1000/mm(3) and a platelet count of 50,000/mm(3) without transfusion.

Patients must have a creatinine of less than 2.0 mg/dL.

Omission of cyotoxic chemotherapy and systemic steroids for 3 weeks prior to entry into the trial is required. Topical and inhaled steroids will be permitted.

Patients must have a life expectancy of greater than 2 months.

Eligible patients must be greater than or equal to 18 years old. There is no upper age limit.

Patients must have SGOT and SGPT value less than or equal to 2.0-fold greater than the upper limit of normal and bilirubin less than or equal to 2.0 mg/dL.

Patients must be able to understand and sign an Informed Consent form.

Karnofsky Performance Status greater than or equal to 70%.

EXCLUSION CRITERIA:

Patients with central nervous system disease as assessed by clinical examination. If the clinical findings suggest the presence of CNS disease a lumbar puncture should be done.

Pregnant and nursing patients are not eligible for the study because the effects of HeFi-1 on the developing fetus and the nursing infant are unknown. All patients must agree to use effective contraceptive measures while receiving therapy and for two weeks afterwards.

HIV positive patients are excluded from the study because the toxicity may be different in this population.

Hepatitis B surface antigen positive and Hepatitis C antibody positive patients are excluded because the toxicity of therapy may be different in this population.

Patients who previously received murine monoclonal antibody therapy are ineligible.

Patients who are HAMA positive.

Patients with significant renal, pulmonary, cardiovascular, endocrine, rheumatologic or allergic disease should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2002-11-05; Primary Completion 2008-07-02 (Actual); Study Completion 2008-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Background] Catane R, Longo DL. Monoclonal antibodies for cancer therapy. Isr J Med Sci. 1988 Sep-Oct;24(9-10):471-6. PMID 3060441
- [Background] Grillo-Lopez AJ, White CA, Varns C, Shen D, Wei A, McClure A, Dallaire BK. Overview of the clinical development of rituximab: first monoclonal antibody approved for the treatment of lymphoma. Semin Oncol. 1999 Oct;26(5 Suppl 14):66-73. PMID 10561020
- [Background] Shak S. Overview of the trastuzumab (Herceptin) anti-HER2 monoclonal antibody clinical program in HER2-overexpressing metastatic breast cancer. Herceptin Multinational Investigator Study Group. Semin Oncol. 1999 Aug;26(4 Suppl 12):71-7. PMID 10482196